CLINICAL TRIAL: NCT00084526
Title: Evaluation of Daily CT Scans Using CT on Rails for Localization in the Treatment of Prostate Cancer
Brief Title: Computed Tomography (CT) Scans Using CT-On-Rails™ to Pinpoint the Location of the Tumor in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000365453; P30CA006927 (NIH); FCCC-03005
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: computed tomography
Procedure: ultrasound imaging

SUMMARY:
RATIONALE: New imaging procedures such as CT-on-rails™ may improve the ability to pinpoint the location of the tumor and decrease radiation therapy damage to healthy tissue.

PURPOSE: This phase I/II trial is studying how well computed tomography (CT) scans using CT-on-rails™ work in pinpointing the location of the tumor in patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Validate the software for CT-on-rails™ by comparing prostate target localization via daily ultrasound vs computed tomography (CT) in patients undergoing radiotherapy for prostate cancer.

Secondary

* Determine the potential benefit of using fiducials in the prostate of patients undergoing daily CT scans and/or ultrasounds for localization.
* Determine the intra- and inter-radiation treatment setup and target position uncertainties, in terms of isocenter coordinates in space, using both the ultrasound and CT scans compared to the coordinates of the isocenter determined at simulation, in these patients.

OUTLINE: This is a pilot study.

* Phase I: Patients undergo computed tomography (CT) using CT-on-rails™ twice weekly. Patients undergo BAT™ ultrasound daily for prostate localization. Patients undergo concurrent daily radiotherapy off study after imaging. After radiotherapy treatment is complete, patients continue to undergo scanning using CT-on-rails™ twice weekly.
* Phase II: Patients undergo local anesthesia and surgical insertion of gold fiducial markers into the prostate. After 1 week, patients undergo a daily CT scan using CT-on-rails™ and bi-weekly BAT™ ultrasound. Patients undergo daily radiotherapy off study after imaging. After radiotherapy treatment is complete, patients continue to undergo scanning using CT-on-rails™ twice weekly.

PROJECTED ACCRUAL: A total of 40 patients (20 per study phase) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of definitive prostate cancer
* Radiotherapy planned as treatment

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-11; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Validity of CT-on-rails software

SECONDARY OUTCOMES:
Efficacy of fiducials
Treatment setup and target position uncertainties

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States